CLINICAL TRIAL: NCT03189511
Title: Short Term Effect of Fluvastatin on Brown Adipose Tissue Thermogenesis and Activity in Humans
Brief Title: Effect of Fluvastatin on Brown Fat Activity
Acronym: FluvaBAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: University of Basel (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: FluvaBAT
Record Dates: First submitted 2017-06-12; First posted 2017-06-16 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Adipose Tissue, Brown; Insulin Resistance; Clinical Trial
Keywords: Brown Adipose Tissue; Brown Fat; Fluvastatin; Prospective Clinical Trial
MeSH Terms: conditions — Insulin Resistance | interventions — Fluvastatin

STUDY DESIGN:
Intervention Model Description: Open-label non-randomized historic control (before-after) trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Volunteers receive calorimetric tests and FDG PET scans pre and post 2 weeks of Fluvastatine.
  Interventions: Drug: Fluvastatin

INTERVENTIONS:
Drug: Fluvastatin — Fluvastatin 40 mg twice daily per mouth for 14 days.
  Other Names: Lescol

SUMMARY:
The purpose of this study is to elucidate the effects of Fluvastatin on brown adipose tissue activity in humans.

DETAILED DESCRIPTION:
Statins, inhibitors of cholesterol biosynthesis, act by inhibiting the enzyme of the mevalonate pathway. Although the clinical benefits of statins are undisputable, they have been shown to increase insulin resistance and incidence of type 2 diabetes mellitus, the mechanism of which is currently not clear.

The main function of brown adipose tissue (BAT) is non-shivering thermogenesis (i.e. heat production through energy dissipation) in brown adipocytes. There has been a growing interest in BAT as a novel therapeutic approach to increase energy expenditure in order to facilitate weight-loss and increase insulin sensitivity.

BAT activity will be assessed using calorimetric test and [18F]-Fluorodeoxyglucose (FDG) positron emission tomography (PET).

We speculate that statins inhibit BAT function and that this mechanism may contribute to the above mentioned increase in insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers (18-40 y)
* body mass index 19 to 27 kg/m²
* Fluent in German or English

Exclusion Criteria:

* Regular physical exercise of more than >150 min of exercise per week.
* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product,
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.),
* Clinically indicated intake of the following medications: Corticosteroids, CYP3A4-Inhibitors (Itraconazol, Voriconazol, Fluconazol, Clarithromycin, Erythromycin, Indinavir, Nelfinavir, Ritonavir, Grapefruit juice), Beta-Blocker, Neuroleptics, Tricyclic Antidepressants,
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Participation in another study involving ionizing radiation in the same year,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons,
* MRI contraindications: Not MRI-compatible metal in the body, cardiac pacemaker, History of surgery with possible metal clips/parts still in the body, claustrophobia.
* Resting pulse rate > 70 bpm
* Known arterial hypertension or resting blood pressure > 130/80 mmHg.
* frequence corrected QT-time (QTc) >430 ms
* Serum creatinine > 1.5x upper limit of norm (ULN), i.e.> 145 µmol/L
* creatine kinase > 1.5x ULN, i.e. > 300 U/L
* aspartate transaminase (ASAT) > 1.5x ULN, i.e. > 51 U/L
* alanine aminotransferase (ALAT) > 1.5x ULN, i.e. > 88 U/L
* Hypothyroidism
* Vitamin D deficiency, Vitamin D3 < 25 nmol/L
* Intake of anticoagulants or inhibitors of platelet aggregation (e.g. Aspirin, clopidogrel).
* Known tendency to form keloids (hypertrophic scar tissue)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-02-19 (Actual)

PRIMARY OUTCOMES:
(18)F-FDG uptake in the supraclavicular brown adipose tissue measured by PET by the maximum standardized uptake value (SUVmax) | 14 days
  Cold and Mirabegron induced 18F-FDG uptake into the supra-clavicular brown adipose tissue (scBAT) as determined by 18F-FDG PET/MR standardized uptake value (SUVmax) after two weeks of treatment with Fluvastatin.

SECONDARY OUTCOMES:
The mean standardized uptake value for 18F-FDG uptake (SUVmean) in the supraclavicular adipose tissue depot | 14 days
  SUVmean in the supraclavicular adipose tissue depot (analog. SUVmax)
Volume of supraclavicular BAT | 14 days
  Volume of supraclavicular BAT as determined on Magnetic Resonance Imaging (MRI)
fat fraction with T2 relaxation time of the BAT depot | 14 days
  fat fraction with T2 relaxation time of the scBAT depot as determined by MRI
Cold induced thermogenesis | 14 days
  Cold induced thermogenesis: Increase in energy expenditure above resting metabolic rate in response to a mild cold stimulus and pharmacologic stimulation with Mirabegron.
Supraclavicular skin temperature in response to mild cold stimulus | 14 days
  Supraclavicular skin temperature in response to mild cold stimulus measured by local probe

CONTACTS AND LOCATIONS:
Overall Officials: Irene A Burger, M.D., Principal Investigator — University of Zurich
Locations (2):
- Switzerland (2):
  - University Hospital of Zurich, PET/MR Center, Schlieren, Canton of Zurich
  - University Hospital of Basel, Basel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cypess AM, Weiner LS, Roberts-Toler C, Franquet Elia E, Kessler SH, Kahn PA, English J, Chatman K, Trauger SA, Doria A, Kolodny GM. Activation of human brown adipose tissue by a beta3-adrenergic receptor agonist. Cell Metab. 2015 Jan 6;21(1):33-8. doi: 10.1016/j.cmet.2014.12.009. PMID 25565203
- [Background] Preiss D, Seshasai SR, Welsh P, Murphy SA, Ho JE, Waters DD, DeMicco DA, Barter P, Cannon CP, Sabatine MS, Braunwald E, Kastelein JJ, de Lemos JA, Blazing MA, Pedersen TR, Tikkanen MJ, Sattar N, Ray KK. Risk of incident diabetes with intensive-dose compared with moderate-dose statin therapy: a meta-analysis. JAMA. 2011 Jun 22;305(24):2556-64. doi: 10.1001/jama.2011.860. PMID 21693744
- [Background] Puurunen J, Piltonen T, Puukka K, Ruokonen A, Savolainen MJ, Bloigu R, Morin-Papunen L, Tapanainen JS. Statin therapy worsens insulin sensitivity in women with polycystic ovary syndrome (PCOS): a prospective, randomized, double-blind, placebo-controlled study. J Clin Endocrinol Metab. 2013 Dec;98(12):4798-807. doi: 10.1210/jc.2013-2674. Epub 2013 Oct 23. PMID 24152688
- [Background] Duvnjak L, Blaslov K. Statin treatment is associated with insulin sensitivity decrease in type 1 diabetes mellitus: A prospective, observational 56-month follow-up study. J Clin Lipidol. 2016 Jul-Aug;10(4):1004-1010. doi: 10.1016/j.jacl.2016.04.012. Epub 2016 May 10. PMID 27578133
- [Background] Chapple CR, Dvorak V, Radziszewski P, Van Kerrebroeck P, Wyndaele JJ, Bosman B, Boerrigter P, Drogendijk T, Ridder A, Van Der Putten-Slob I, Yamaguchi O; Dragon Investigator Group. A phase II dose-ranging study of mirabegron in patients with overactive bladder. Int Urogynecol J. 2013 Sep;24(9):1447-58. doi: 10.1007/s00192-013-2042-x. Epub 2013 Mar 8. PMID 23471546
- [Derived] Loeliger RC, Maushart CI, Gashi G, Senn JR, Felder M, Becker AS, Muller J, Balaz M, Wolfrum C, Burger IA, Betz MJ. Relation of diet-induced thermogenesis to brown adipose tissue activity in healthy men. Am J Physiol Endocrinol Metab. 2021 Jan 1;320(1):E93-E101. doi: 10.1152/ajpendo.00237.2020. Epub 2020 Nov 23. PMID 33225717
- [Derived] Fischer JGW, Maushart CI, Becker AS, Muller J, Madoerin P, Chirindel A, Wild D, Ter Voert EEGW, Bieri O, Burger I, Betz MJ. Comparison of [18F]FDG PET/CT with magnetic resonance imaging for the assessment of human brown adipose tissue activity. EJNMMI Res. 2020 Jul 22;10(1):85. doi: 10.1186/s13550-020-00665-7. PMID 32699996